CLINICAL TRIAL: NCT06275139
Title: Integrated Assessment of Cervicocerebral Vessels by Multidisciplinary Team to Improve the Brain Injury for CAGB Patients With High Risk of Stroke (IACV Study)
Brief Title: Integrated Assessment of Cervicocerebral Vessels to Improve the Brain Injury for CAGB Patients (IACV Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-GSP-GG-9
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronary Disease; Coronary Artery Bypass; Strokes Thrombotic
Keywords: Coronary Disease; Coronary artery bypass; Stroke
MeSH Terms: conditions — Coronary Disease; Thrombotic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Integrated assessment of cervicocerebral vessels shall be performed, including transcranial color-coded doppler, cerebral perfusion with multislice CT, and cognitive function assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No-integrated group) (No Intervention): The control group adopt the traditional diagnosis and treatment mode, and only head CT plain scan and carotid artery ultrasound shall be performed. If necessary, relevant disciplines would be consulted but no integrated assessment of cervicocerebral vessels be arranged. The final treatment plan would be decided by the surgeon alone.
- Experimental group (Integrated group) (Experimental): The experimental group adopt the multidisciplinary collaboration and integrated evaluation mode. In addition to routine diagnosis and treatment as above-mentioned, integrated assessment of cervicocerebral vessels shall be performed, including transcranial color-coded doppler, cerebral perfusion with multislice CT, and cognitive function assessment. Based on the above results, surgical plans will be formulated jointly by multiple disciplines including neurologists, vascular surgeons, ICU physicians and cardiac surgeons.
  Interventions: Other: Integrated Assessment of Cervicocerebral Vessels

INTERVENTIONS:
Other: Integrated Assessment of Cervicocerebral Vessels — Integrated assessment of cervicocerebral vessels shall be performed, including transcranial color-coded doppler, cerebral perfusion with multislice CT, and cognitive function assessment.
  Arms: Experimental group (Integrated group)

SUMMARY:
The goal of this study is to establish a prospective study to focus on the high-risk stroke population who require coronary artery bypass graft surgery. It will divide the eligible patients into 1:1 group by simple randomization method. The control group adopt the traditional diagnosis and treatment mode, and only head CT plain scan and carotid artery ultrasound shall be performed. If necessary, relevant disciplines would be consulted but no integrated assessment of cervicocerebral vessels be arranged. The final treatment plan would be decided by the surgeon alone. The experimental group adopt the multidisciplinary collaboration and integrated evaluation mode. In addition to routine diagnosis and treatment as above-mentioned, integrated assessment of cervicocerebral vessels shall be performed, including transcranial color-coded doppler, cerebral perfusion with multislice CT, and cognitive function assessment. Based on the above results, surgical plans will be formulated jointly by multiple disciplines including neurologists, vascular surgeons, ICU physicians and cardiac surgeons. Researchers will compare the two groups to investigate whether integrated assessment of cervicocerebral vessels can reduce the incidence of brain injury compared with conventional diagnosis and treatment mode.

DETAILED DESCRIPTION:
Brain injury is one of the most important factors leading to poor prognosis of CABG surgery, especially for high-risk patients. In order to reduce brain injury after cardiac surgery, preoperative assessment and management are particularly important. Multidisciplinary diagnosis and treatment mode (multidisciplinary team, MDT) refers to a multidisciplinary clinical work team, usually a fixed working group composed of several related disciplines. MDT carries out routine clinical discussions for difficult and complex disease and develop accurate and effective individualized treatment plans for patients, which has become the mainstream trend. The traditional treatment mode mainly relies on head CT and carotid ultrasound to evaluate the nervous system, and then the surgeon decides the operation mode according to experience, ignoring the role of related disciplines, including neurologists, vascular surgeons, ICU physicians and cardiac surgeons. We believe that integrated assessment of cervicocerebral vessels will help reduce the incidence of brain injury in high-risk patients. This study is an exploratory attempt for high-risk patients, which can provide more evidence for the prevention of perioperative neurological complications of CABG, and is of great significance for reducing disease burden, ensuring surgical safety, and improving the long-term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require CABG surgery; Age ≥18 years with a history of stroke or transient ischemic attack; Combined with typical symptoms of stroke; Previous imaging findings suggest a high risk of stroke

Exclusion Criteria:

* < 18 years old; > 80 years old; Combined with congenital cerebrovascular malformation; Emergency operation; Reluctant to sign an informed consent form; Reluctant to follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of neurological complications | Within three months after surgery
  Diagnosed by clinical manifestation, brain CT or MRI

SECONDARY OUTCOMES:
The incidence of major adverse cardiac events | Within three months after surgery
  Diagnosed by follow up
Neurological scale scores | Within 3 months after surgery
  Measured by using neurological system scale

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Fuwai Hospital; National Cardiovascular Center
Locations (1):
- Fuwai Hospital; National Cardiovascular Center; Peking Union Medical College & Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ottens TH, Dieleman JM, Sauer AM, Peelen LM, Nierich AP, de Groot WJ, Nathoe HM, Buijsrogge MP, Kalkman CJ, van Dijk D; DExamethasone for Cardiac Surgery (DECS) Study Group. Effects of dexamethasone on cognitive decline after cardiac surgery: a randomized clinical trial. Anesthesiology. 2014 Sep;121(3):492-500. doi: 10.1097/ALN.0000000000000336. PMID 25225745
- [Result] Greaves D, Psaltis PJ, Davis DHJ, Ross TJ, Ghezzi ES, Lampit A, Smith AE, Keage HAD. Risk Factors for Delirium and Cognitive Decline Following Coronary Artery Bypass Grafting Surgery: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2020 Nov 17;9(22):e017275. doi: 10.1161/JAHA.120.017275. Epub 2020 Nov 7. PMID 33164631
- [Result] Kumpaitiene B, Svagzdiene M, Sirvinskas E, Adomaitiene V, Petkus V, Zakelis R, Krakauskaite S, Chomskis R, Ragauskas A, Benetis R. Cerebrovascular autoregulation impairments during cardiac surgery with cardiopulmonary bypass are related to postoperative cognitive deterioration: prospective observational study. Minerva Anestesiol. 2019 Jun;85(6):594-603. doi: 10.23736/S0375-9393.18.12358-3. Epub 2018 May 11. PMID 29756691
- [Result] Leenders J, Overdevest E, van Straten B, Golab H. The influence of oxygen delivery during cardiopulmonary bypass on the incidence of delirium in CABG patients; a retrospective study. Perfusion. 2018 Nov;33(8):656-662. doi: 10.1177/0267659118783104. Epub 2018 Jun 29. PMID 29956559
- [Result] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936
- [Result] Yilmaz S, Aksoy E, Diken AI, Yalcinkaya A, Erol ME, Cagli K. Dopamine Administration is a Risk Factor for Delirium in Patients Undergoing Coronary Artery Bypass Surgery. Heart Lung Circ. 2016 May;25(5):493-8. doi: 10.1016/j.hlc.2015.09.012. Epub 2015 Oct 22. PMID 26546094
- [Result] Crocker E, Beggs T, Hassan A, Denault A, Lamarche Y, Bagshaw S, Elmi-Sarabi M, Hiebert B, Macdonald K, Giles-Smith L, Tangri N, Arora RC. Long-Term Effects of Postoperative Delirium in Patients Undergoing Cardiac Operation: A Systematic Review. Ann Thorac Surg. 2016 Oct;102(4):1391-9. doi: 10.1016/j.athoracsur.2016.04.071. Epub 2016 Jun 22. PMID 27344279
- [Result] Eide LS, Ranhoff AH, Fridlund B, Haaverstad R, Hufthammer KO, Kuiper KK, Nordrehaug JE, Norekval TM; CARDELIR Investigators. Comparison of frequency, risk factors, and time course of postoperative delirium in octogenarians after transcatheter aortic valve implantation versus surgical aortic valve replacement. Am J Cardiol. 2015 Mar 15;115(6):802-9. doi: 10.1016/j.amjcard.2014.12.043. Epub 2015 Jan 6. PMID 25644851
- [Result] Colak Z, Borojevic M, Bogovic A, Ivancan V, Biocina B, Majeric-Kogler V. Influence of intraoperative cerebral oximetry monitoring on neurocognitive function after coronary artery bypass surgery: a randomized, prospective study. Eur J Cardiothorac Surg. 2015 Mar;47(3):447-54. doi: 10.1093/ejcts/ezu193. Epub 2014 May 7. PMID 24810757
- [Result] van Meenen LC, van Meenen DM, de Rooij SE, ter Riet G. Risk prediction models for postoperative delirium: a systematic review and meta-analysis. J Am Geriatr Soc. 2014 Dec;62(12):2383-90. doi: 10.1111/jgs.13138. PMID 25516034
- [Result] Palmbergen WA, van Sonderen A, Keyhan-Falsafi AM, Keunen RW, Wolterbeek R. Improved perioperative neurological monitoring of coronary artery bypass graft patients reduces the incidence of postoperative delirium: the Haga Brain Care Strategy. Interact Cardiovasc Thorac Surg. 2012 Oct;15(4):671-7. doi: 10.1093/icvts/ivs317. Epub 2012 Jul 9. PMID 22778141
- [Result] Siepe M, Pfeiffer T, Gieringer A, Zemann S, Benk C, Schlensak C, Beyersdorf F. Increased systemic perfusion pressure during cardiopulmonary bypass is associated with less early postoperative cognitive dysfunction and delirium. Eur J Cardiothorac Surg. 2011 Jul;40(1):200-7. doi: 10.1016/j.ejcts.2010.11.024. Epub 2010 Dec 18. PMID 21168339
- [Result] Liu YH, Wang DX, Li LH, Wu XM, Shan GJ, Su Y, Li J, Yu QJ, Shi CX, Huang YN, Sun W. The effects of cardiopulmonary bypass on the number of cerebral microemboli and the incidence of cognitive dysfunction after coronary artery bypass graft surgery. Anesth Analg. 2009 Oct;109(4):1013-22. doi: 10.1213/ane.0b013e3181aed2bb. PMID 19762724
- [Result] Scott DA, Silbert BS, Doyle TJ, Blyth C, Borton MC, O'brien JL, de L Horne DJ. Centrifugal versus roller head pumps for cardiopulmonary bypass: effect on early neuropsychologic outcomes after coronary artery surgery. J Cardiothorac Vasc Anesth. 2002 Dec;16(6):715-22. doi: 10.1053/jcan.2002.128413. PMID 12486652
- [Result] Harmon DC, Ghori KG, Eustace NP, O'Callaghan SJ, O'Donnell AP, Shorten GD. Aprotinin decreases the incidence of cognitive deficit following CABG and cardiopulmonary bypass: a pilot randomized controlled study. Can J Anaesth. 2004 Dec;51(10):1002-9. doi: 10.1007/BF03018488. PMID 15574551
- [Result] Marijon E, Narayanan K, Smith K, Barra S, Basso C, Blom MT, Crotti L, D'Avila A, Deo R, Dumas F, Dzudie A, Farrugia A, Greeley K, Hindricks G, Hua W, Ingles J, Iwami T, Junttila J, Koster RW, Le Polain De Waroux JB, Olasveengen TM, Ong MEH, Papadakis M, Sasson C, Shin SD, Tse HF, Tseng Z, Van Der Werf C, Folke F, Albert CM, Winkel BG. The Lancet Commission to reduce the global burden of sudden cardiac death: a call for multidisciplinary action. Lancet. 2023 Sep 9;402(10405):883-936. doi: 10.1016/S0140-6736(23)00875-9. Epub 2023 Aug 27. PMID 37647926
- [Result] Izzy M, Fortune BE, Serper M, Bhave N, deLemos A, Gallegos-Orozco JF, Guerrero-Miranda C, Hall S, Harinstein ME, Karas MG, Kriss M, Lim N, Palardy M, Sawinski D, Schonfeld E, Seetharam A, Sharma P, Tallaj J, Dadhania DM, VanWagner LB. Management of cardiac diseases in liver transplant recipients: Comprehensive review and multidisciplinary practice-based recommendations. Am J Transplant. 2022 Dec;22(12):2740-2758. doi: 10.1111/ajt.17049. Epub 2022 Apr 22. PMID 35359027